CLINICAL TRIAL: NCT01752517
Title: A Phase Ⅱ Single-arm Clinical Trial to Investigate the Efficacy and Safety of Vinorelbine-ifosfamide Regimen as Third-line Treatment in Refractory or Recurrent Extensive Small Cell Lung Cancer Patients
Brief Title: Vinorelbine and Ifosfamide as Third-line Treatment for Refractory Small Cell Lung Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PUMCH-S463
Record Dates: First submitted 2012-12-12; First posted 2012-12-19 (Estimated); Last update posted 2012-12-19 (Estimated); Status verified 2012-12

CONDITIONS: Small Cell Lung Cancer
Keywords: small cell lung cancer; chemotherapy; vinorelbine; ifosfamide; third-line treatment
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Vinorelbine; Ifosfamide; Mesna

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- refractory SCLC: NI group vinorelbine 25mg/m2 d1,d8; Ifosfamide 1.25g/m2 d1-d3; Mesna 400mg iv 0,4,8 hours after ifosfamide administration for 3 days; every 3 weeks; up to the maximum cycles (total:6);
  Interventions: Drug: NI group

INTERVENTIONS:
Drug: NI group — vinorelbine 25mg/m2 d1,d8; ifosfamide 1.25g/m2 d1-d3; Mesna 400mg iv 0,4,8 hours after ifosfamide administration for 3 days
  Other Names: vinorelbine;; ifosfamide;; Mesna;

SUMMARY:
Although fist-line therapy with Cisplatin and etoposide(EP)or Carboplatin and etoposide(CE)and second-line therapy with topotecan has been given, patients with ED-SCLC still relapse and 2-year survival is less than 10%. There is no standard treatment recommendation for this group of patients who failed to second-line therapy and had good performance status. Some cytotoxic drugs for the treatment of non-small cell lung cancer, i.e. vinorelbine, paclitaxel, and ifosfamide, were used in refractory or recurrent SCLC patients. Recently, a retrospective study showed the overall response rate was 30%, the median progression free survival (PFS) was 6.5 months, and the median overall survival was 10.4 months in advanced combined SCLC patients treated with first-line regimen of vinorelbine, ifosfamide and cisplatin (NIP). Because of the previous platinum administration and patient's performance status, only vinorelbine and ifosfamide (NI) are combined and used as third-line therapy for refractor or recurrent ED-SCLC in our lung cancer center. And this clinical trial is designed to prospectively investigate the efficacy and safety of NI regimen in refractory or recurrent ED-SCLC patients in our center.

DETAILED DESCRIPTION:
Small cell lung cancer (SCLC) is a highly aggressive disease characterized by its rapid doubling time, high growth fraction, early development of disseminated disease, and dramatic response to first-line chemotherapy and radiation. Small cell lung cancer accounts for approximately 20%-25% lung cancer patients. SCLC patients are categorized as limited disease, defined as disease that is confined to the ipsilateral hemithorax that can be encompassed within a tolerable radiation port, or extensive disease (ED), defined as the presence of overt metastatic disease determined by imaging or physical examination. Two third of patients are diagnosed with ED at presentation. Despite the development of novel cytotoxic drugs, the therapeutic approach to SCLC has been stagnant for more than twenty years. Standard treatment for ED-SCLC remains EP or CE, a regimen that yield a median survival of approximately 9 months and a 5-year survival of less than 1%.

Most patients are destined to relapse, and the prognosis for this group of patients who relapse is poor. Patients who relapse < 3 months after first-line therapy are commonly called refractory, and patients who relapse 3 months after therapy are labeled as sensitive. In a randomized multicenter study, von Pawel et al compared cyclophosphamide, adriamycin, and vincristine (CAV) with topotecan as a single agent in patients who had relapse at least 60 days (2 months) after initial therapy. The response rates were 24.3% in patients treated with topotecan and 18.3% in patients treated with CAV (P=0.285). Median times to progression were 13.3 weeks for the topotecan arm and 12.3 weeks for the CAV arm. Median survival times were 25 weeks for topotecan and 24.7 weeks for CAV. The proportion of patients with symptom improvement was greater in the topotecan arm than in the CAV arm. The authors concluded that topotecan was at least as effective as CAV in the treatment of patients with recurrent SCLC. So in some guidelines for SCLC, topotecan is recommended as the standard second-line treatment in patients who relapse less than 3 months. As for patients who relapse more than six months after the end of initial treatment, EP or CE regimen is recommended to be used again.

ELIGIBILITY:
Inclusion Criteria:

* histologically or cytologically confirmed ED-SCLC;
* age>18 and <75;
* measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST);
* previous treatments including first-line therapy with EP or CE and second-line therapy with topotecan;
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-2;
* life expectancy > 3 months;
* neutrophil count > 1500/ul;
* platelet count > 100,000ul;
* hemoglobin level > 9g/dl;
* bilirubin level < 1.5mg/dL;
* creatinine level < 2mg/dl;
* alanine transaminase (AST) levels < 2.5× upper limit of normal (ULN)(or < 5× ULN if liver metastases were present);

Exclusion Criteria:

* previous anticancer therapy including vinorelbine or ifosfamide;
* newly diagnosed central nervous system (CNS) metastasis and not treated by radiotherapy or surgery;
* additional malignancies;
* uncontrolled systemic disease;
* pregnancy or breast feeding phase;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ED-SCLC patients who relapse after treatment with first-line EP or CE and second-line topotecan.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2012-12; Primary Completion 2014-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
the disease control rate | up to 9 weeks
  The disease control rate includes the rate of progression disease,partial remission and stable disease.

SECONDARY OUTCOMES:
progression free survival | up to 52 weeks (about one year)
  From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 52 weeks.
Overall survival | Up to 100 weeks
  From date of randomization until the date of death from any cause, assessed up to 100 weeks.
the score of functional assessment of cancer treatment-lung (FACT-L) | up to 52 weeks
  FACT-L ia assessed at different time points. (Date of randomization, 1 weeks after chemotherapy, every cycle of chemotherapy, every month after chemotherapy,up to 52 weeks)
Number of participants with adverse events | Up to six months
  The adverse events are assessed by National Cancer Institute-Common Toxicity Criteria (Version 3.0)(NCI-CTC).

CONTACTS AND LOCATIONS:
Overall Officials: Mengzhao Wang, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Department of Respiratory Medicine, Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Result] Jackman DM, Johnson BE. Small-cell lung cancer. Lancet. 2005 Oct 15-21;366(9494):1385-96. doi: 10.1016/S0140-6736(05)67569-1. PMID 16226617
- [Result] Simon GR, Turrisi A; American College of Chest Physicians. Management of small cell lung cancer: ACCP evidence-based clinical practice guidelines (2nd edition). Chest. 2007 Sep;132(3 Suppl):324S-339S. doi: 10.1378/chest.07-1385. PMID 17873178
- [Result] Clark R, Ihde DC. Small-cell lung cancer: treatment progress and prospects. Oncology (Williston Park). 1998 May;12(5):647-58; discussion 661-3. PMID 9597676
- [Result] Fukuoka M, Furuse K, Saijo N, Nishiwaki Y, Ikegami H, Tamura T, Shimoyama M, Suemasu K. Randomized trial of cyclophosphamide, doxorubicin, and vincristine versus cisplatin and etoposide versus alternation of these regimens in small-cell lung cancer. J Natl Cancer Inst. 1991 Jun 19;83(12):855-61. doi: 10.1093/jnci/83.12.855. PMID 1648142
- [Result] Wolf M, Havemann K, Holle R, Gropp C, Drings P, Hans K, Schroeder M, Heim M, Dommes M, Mende S, et al. Cisplatin/etoposide versus ifosfamide/etoposide combination chemotherapy in small-cell lung cancer: a multicenter German randomized trial. J Clin Oncol. 1987 Dec;5(12):1880-9. doi: 10.1200/JCO.1987.5.12.1880. PMID 2824710
- [Result] Roth BJ, Johnson DH, Einhorn LH, Schacter LP, Cherng NC, Cohen HJ, Crawford J, Randolph JA, Goodlow JL, Broun GO, et al. Randomized study of cyclophosphamide, doxorubicin, and vincristine versus etoposide and cisplatin versus alternation of these two regimens in extensive small-cell lung cancer: a phase III trial of the Southeastern Cancer Study Group. J Clin Oncol. 1992 Feb;10(2):282-91. doi: 10.1200/JCO.1992.10.2.282. PMID 1310103
- [Result] Skarlos DV, Samantas E, Kosmidis P, Fountzilas G, Angelidou M, Palamidas P, Mylonakis N, Provata A, Papadakis E, Klouvas G, et al. Randomized comparison of etoposide-cisplatin vs. etoposide-carboplatin and irradiation in small-cell lung cancer. A Hellenic Co-operative Oncology Group study. Ann Oncol. 1994 Sep;5(7):601-7. doi: 10.1093/oxfordjournals.annonc.a058931. PMID 7993835
- [Result] von Pawel J, Schiller JH, Shepherd FA, Fields SZ, Kleisbauer JP, Chrysson NG, Stewart DJ, Clark PI, Palmer MC, Depierre A, Carmichael J, Krebs JB, Ross G, Lane SR, Gralla R. Topotecan versus cyclophosphamide, doxorubicin, and vincristine for the treatment of recurrent small-cell lung cancer. J Clin Oncol. 1999 Feb;17(2):658-67. doi: 10.1200/JCO.1999.17.2.658. PMID 10080612
- [Result] Luo J, Wu FY, Li AW, Zheng D, Liu JM. Comparison of vinorelbine, ifosfamide and cisplatin (NIP) and etoposide and cisplatin (EP) for treatment of advanced combined small cell lung cancer (cSCLC) patients: a retrospective study. Asian Pac J Cancer Prev. 2012;13(9):4703-6. doi: 10.7314/apjcp.2012.13.9.4703. PMID 23167406